CLINICAL TRIAL: NCT06308562
Title: A Pilot Study of Fuzzy Wale Compression Stockinet to Evaluate Healing Following Transtibial Amputation for Peripheral Arterial Disease
Brief Title: Fuzzy Wale Compression Stockinet to Promote Healing Following Transtibial Amputation for Peripheral Arterial Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Matthew M. Melin, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-010717
Record Dates: First submitted 2024-03-07; First posted 2024-03-13 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Fuzzy Wale Compression Stockinet (Experimental): Subjects with peripheral arterial disease requiring transtibial amputation will have Fuzzy Wale Compression Stockinet applied and utilized for 4-8 weeks post operatively or until prosthetic fitting and wound has achieved full durable healing.
  Interventions: Device: Fuzzy Wale Compression Stockinet
- Standard of care (No Intervention): Subjects with peripheral arterial disease requiring transtibial amputation will receive standard of care treatment compression stockinet.

INTERVENTIONS:
Device: Fuzzy Wale Compression Stockinet — EdemaWear is a tubular, circular knit elastic stockinet fabricated with elastic, vertically oriented fuzzy wales, with the compression provided by the elastic, horizontal oriented Lycra® spandex yarns knitted in between. The stockinet is applied from the foot to the popliteal crease, over the affected area. EdemaWear can be applied in direct contact with the skin or over a wound care dressing. Sizing is based on leg circumference. EdemaWear is indicated for edema management of various etiologies (lymphedema, chronic venous insufficiency, congestive heart failure), and optimizing wound healing. The stockinette is often combined with other boxed compression sets. The manufacturer's stated dosage of EdemaWear is 8-12mmHg when used alone.
  Other Names: EdemaWear
  Arms: Fuzzy Wale Compression Stockinet

SUMMARY:
The objective of this study is to determine if using Fuzzy Wale compression stockinet can assist in reducing the healing time and decrease costs in transtibial amputation patients as compared to standard of care treatment compression stocking.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* Male and female
* Transtibial amputation expected.
* Peripheral arterial disease and Transcutaneous partial pressure of oxygen (TCP02, if performed)
* Ability of subject to give appropriate consent or have an appropriate representative available to do so.

Exclusion Criteria:

* Known allergies to any of the components of the compression.
* Terminal illness or current cancer therapy with chemotherapy
* Inability to undergo ongoing care in Rochester.
* Lack of cognitive ability to follow instructions or monitor residual limb.
* Vulnerable study population
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Surgical site infection | 8 weeks post-operatively
  Number of subject presenting with surgical site infections following transtibial amputation.
Wound dehiscence | 8 weeks post-operatively
  Number of subject presenting with wound dehiscence following transtibial amputation.
Pain control | 8 weeks post-operatively
  Pain control during healing following transtibial amputation will be measured using the Visual Analog Scale (VAS). VAS scores range from 0-10 with 10 being the worst possible pain and 0 being no pain.
Time to prosthetic fitting | 8 weeks post-operatively
  Number of days from transtibial amputation to prosthetic fitting.

SECONDARY OUTCOMES:
Length of hospital stay | 8 weeks post-operatively
  Number of days from transtibial amputation to hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Melin, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No